CLINICAL TRIAL: NCT07281482
Title: Randomised Controlled Trial of a Cognitive, Emotional and Social Stimulation Programme for Socioeconomically Disadvantaged Children.
Brief Title: Study Protocol: Cognitive, Emotional and Social Stimulation Programme for Low-SES Children.
Acronym: Activa-Mente
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Joan Deus Yela (Other)
Collaborators: Cognifit (Unknown); Universitat Autonoma de Barcelona (Other); Universidad Loyola Andalucia (Other); Universidad de San Buenaventura (Other); Neuronup S.L. (Unknown)
Responsible Party: Sponsor-Investigator, Joan Deus Yela, Doctor en Psicología, Universitat Autonoma de Barcelona
Organization: Universitat Autonoma de Barcelona (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: UAB-ACTIVA-MENTE-2025-01
Record Dates: First submitted 2025-11-19; First posted 2025-12-15 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-10

CONDITIONS: Child Development; Socioeconomic Factors
Keywords: cognitive stimulation; vulnerability; child development; Neuropsychology; Emotional stimulation; randomized controlled trials

STUDY DESIGN:
Intervention Model Description: This research will employ a cluster randomised controlled trial design, as the class or school group receiving the intervention will be randomly selected and compared with another group engaged in regular educational activities conducted concurrently. The study will be conducted in real contexts, and schools will be invited to participate through an open call. Participants will be randomly assigned per class group to the experimental group, while the remaining participants will constitute the control group. The intervention programme will be offered to all participating children in the class that is part of the experimental group. The research team will ensure that both groups are homogeneous in their demographic characteristics (age, gender, socioeconomic status).
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive stimulation group (Experimental): The experimental group receives cognitive stimulation through platforms such as Cognifit and Neuronup.
  Interventions: Other: Cognitive and emotional stimulation; Behavioral: Training for parents and teachers
- placebo group (Placebo Comparator): The control group receives random activities that do not affect their cognitive development.
  Interventions: Other: Random activities

INTERVENTIONS:
Other: Cognitive and emotional stimulation — Continuous cognitive and emotional stimulation is provided in the school setting.
  Arms: Cognitive stimulation group
Other: Random activities — Random activities will be carried out for the control group that will not include the improvement of cognitive functions.
  Arms: placebo group
Behavioral: Training for parents and teachers — Training in neuroeducation and learning strategies focused on brain function will be provided for teachers and parents, with the level of depth appropriate for each group.
  Arms: Cognitive stimulation group

SUMMARY:
Latin America and the Caribbean exhibit high rates of poverty and social exclusion, where a significant portion of the population faces challenges in meeting basic needs. This socioeconomic vulnerability exacerbates environmental violence and its associated consequences. Recognizing that contexts of poverty and social exclusion can adversely impact children's cognitive and emotional development, this research protocol aims to address these challenges. It proposes a cognitive and emotional stimulation program, complemented by an intervention targeting teachers and caregivers, grounded in neuroeducational principles. The overarching goal is to enhance children's cognitive and academic performance, thereby improving their long-term quality of life. Methods: A randomised controlled trial will be conducted to evaluate the efficacy of the intervention in an experimental group compared to a control group. A sample of more than 500 children from primary schools in disadvantaged contexts in Colombia A digital stimulation programme, designed and supervised by neuropsychologists, will be implemented within the classrooms and will be complemented with educational sessions in neuroeducation for teachers and caregivers, with weekly activities for 3 months. Three evaluations will be carried out: 1) pre-intervention, 2) post-intervention and 3) follow-up. During follow-up, the control group will receive the stimulation programme. Conclusions: The researchers anticipate a positive impact on the cognitive, emotional and academic performance of these children, providing evidence and support for the long-term creation of a tested and validated cognitive and emotional stimulation programme that could be integrated into the academic curriculum of educational centres in disadvantaged contexts.

DETAILED DESCRIPTION:
There is evidence of a large gap in the cognitive development of children and adolescents in violent contexts and situations of socio-economic vulnerability. There are multiple reasons that affect the cognitive and emotional development of these children, who are at a disadvantage with respect to children of the same age who are not in the same situation or who enjoy better contextual situations. Poor nutrition, the type of stimulation provided by the environment, stressful situations and the constant subjection of the brain to states of alertness encourage the deficiencies found in their integral development. This neuropsychological stimulation programme specifically designed for children at risk of social exclusion aims to be an effective tool in strengthening some of the cognitive abilities with the greatest evidence of impairment, in this case, language (e.g., vocabulary, comprehension and expression), attention (especially the ability to sustain it voluntarily for prolonged periods of time: concentration), and executive functions (set of skills that allow us to voluntarily regulate our behaviour thanks to the inhibition of responses, planning, reasoning and flexible decision making adjusted to the demands of the environment).

In response to the results and observations of the studies carried out within the framework of project 0C138/2020 'MEJORA GUATE', this research proposes intervention objectives for the needs of the participating population, based on a more holistic strategy that integrates the child and their immediate environment. Considering that caregivers and teachers mediate cognitive, emotional, and social development, this project seeks to improve the impact on the different areas of the child's performance. To achieve the planned objectives, work will be carried out through three main axes of application: the neuropsychological stimulation axis, the neurodevelopment training axis, and the dissemination axis, which will in turn be divided into two phases.

The Neuropsychological Stimulation Axis: aims to improve and enhance the development of the cognitive and emotional skills of children from disadvantaged areas of Colombia through direct intervention with them through group activities carried out in their usual educational contexts. To this end, innovative neuropsychological tools from the clinical care of children with neurodevelopmental disorders will be applied to the cognitive and emotional stimulation of these children at risk of social exclusion.

The Training Axis: will build the knowledge base on neurodevelopment and brain function in learning, with the aim of promoting best practice in the implementation of teaching staff, as well as parenting practices and home support by carers. The training will be delivered in a dual format, face-to-face and online, following pedagogical processes with established didactic objectives, evaluation criteria and monitoring of the training received.

The Dissemination Axis: aims to disseminate the advances and results of the research, as well as the pedagogical content of the training, which will generate a greater social reach by promoting complementary channels through which the content on learning and its brain functioning can be shared with different social actors in a didactic and pedagogical way. In terms of resources, it is proposed to create a handbook of good practices to serve as a model for other educational communities, a website with didactic resources and asynchronous training processes, as well as fluid channels for sharing knowledge through social networks commonly used by these groups, such as WhatsApp or Instagram.

The methodology proposed for the implementation of this project aims to promote, from a didactic, longitudinal and cumulative perspective, the improvement of the academic performance and quality of life of Colombian children at risk of social exclusion. By combining the three axes mentioned above, the researchers hope to achieve long-term improvements in the performance of these children. It is clear to us that a professional who understands how to use children's learning to improve their academic performance and quality of life will not only benefit the children, but also many others who may subsequently benefit from the learning of the teachers and carers involved in the project.

A teacher who understands how their students' brains work can improve their teaching strategies by enhancing learning resources. And a caregiver who recognises and identifies the needs of children's brains when they are learning or reviewing academic content in the home can help them learn more effectively.

Therefore, this proposal aims to strengthen the affected cognitive functions and prevent the persistence of their negative effects on participants. To achieve this latter goal, a contextual intervention is proposed to inform about brain functioning during learning acquisition, addressing key concepts of neurodevelopment and the neurocognitive processes involved in learning. Likewise, it seeks to offer specific strategies to parents, caregivers, and teachers in order to promote critical reflection on the quality of support provided to children. It is hoped that this intervention will not only have a positive impact on educational and care practices during the implementation of the project but also generate sustainable changes over time.

The inclusion of caregivers and teachers in the intervention is based on the analysis of results obtained in previous studies, which show that their participation is key to enhancing the positive effects on children. This measure responds to the need to address contextual factors that, in the absence of adequate support, can limit the effectiveness of interventions aimed exclusively at children.

This cognitive stimulation programme incorporates specific activities that promote emotional intelligence, the ability to recognise emotions (our own and those of others) and social cognition (a set of skills that allow us to understand the thoughts and emotions of others, "putting ourselves in the other person's shoes", thus improving empathy). Consequently, it is expected that the improvement of cognitive and emotional skills will have a positive impact on students' academic performance as one of the basic pillars on which meaningful and lasting learning is based.

In the long term, cognitive, emotional and academic improvements are expected to have a positive effect on the expectations and quality of life of these children at risk of social exclusion. The promotion of comprehensive health and well-being conditions is expected to lead to a more inclusive childhood and social development that will bring them closer to a more hopeful future as adults. Among the innovative elements, the use of web-based neurorehabilitation platforms and digital applications stands out, which until now have only been applied in clinical treatment contexts (neurodevelopmental disorders such as Attention Deficit Hyperactivity Disorder, Intellectual Disability or Autism Spectrum Disorder).

In this project, these tools are made available free of charge to children at risk of social exclusion.

For its part, developing training for educators and caregivers allows the approach from the different contexts involved in the child's learning. These trainings will be face-to-face and online and will rely on the use of new information technologies, video tutorials through social networks, to maximise the participation of educators from different locations and caregivers who usually have limited availability. Overall, these innovations are expected to promote a healthier and more effective environment for children's cognitive and emotional development, with a positive impact on the participants' academic performance, on their quality of life and on the people (teachers and caregivers) who directly or indirectly contribute to it.

ELIGIBILITY:
Inclusion Criteria:

* Child's age (must be enrolled between the fourth and fifth grades of basic primary school and sixth and seventh grades of basic secondary school ).
* Belonging to a school in a disadvantaged area of the city of application.
* Informed consent signed by the participant's legal guardian.
* Verbal consent of the participants.
* Possess basic reading skills in Spanish and sufficient motor skills to handle tablets or use a computer mouse.

Exclusion Criteria:

* Not having basic reading skills in Spanish.
* Being enrolled in a school year other than fourth and fifth grade of elementary school or sixth and seventh grade of secondary school.
* Not belonging to a disadvantaged area of the city of Cali.
* Having a physical disability that prevents the use of tablets and mice.
* Not having signed the participation consent form by their parents.

Ages: 9 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 500 (Estimated)
Dates: Start 2026-01-26 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-01-30 (Estimated)

PRIMARY OUTCOMES:
Pre- and post-intervention scores on the general cognitive assessment battery of Cognifit | 12 months
  The Cognitive Assessment Battery (CAB) studies brain function and performs a comprehensive cognitive screening. It accurately assesses a wide range of skills and detects cognitive well-being (high-medium-low). It identifies weaknesses and strengths in the areas of memory, attention-concentration, executive functions, planning, and coordination. All cognitive scores are classified from 0 to 100. In the case of individual cognitive abilities, this score corresponds to a percentile division of the data into equal groups. In the case of cognitive areas and the overall score, this result corresponds to the average of the scores for individual abilities.
  In all cases, the score is interpreted as follows:
  0-25: cognitive weaknesses. 26-50: expected average range, but below average. 51-75: adequate, above average but within the expected range. 76-100: high, well above what is expected for age and gender.
Pre- and post-intervention scores on the Emotional Intelligence Assessment Battery | 12 months
  The evaluation of emotional skills or emotional intelligence will be carried out by applying the adaptation and standardization of the BarOn Emotional Intelligence Inventory ICE: NA, in children and adolescents. It is an instrument that measures the skills and competencies characteristic of emotional intelligence (ability to understand oneself and others, ability to relate to peers and family members and ability to adapt to the demands of the environment), integrates interpersonal, intrapersonal, stress management, adaptability and mood scales in general. It provides information about the emotional and social intelligence of the person being evaluated.
  Interpretation of scores:
  ≥130: Atypically high emotional and social skills, excellent development. 120-129: Very high, very well developed. 110-119: High, well developed. 90-109: Adequate, average level. 80-89: Low, poorly developed, require improvement. 70-79: Very low, need considerable improvement.
  ≤69: Atypical and deficient.

SECONDARY OUTCOMES:
Pre- and post-intervention scores on the Nonverbal intelligence. TONI 4 | 12 months
  The TONI-4 will be used to assess nonverbal intelligence. This test is administered individually to people aged 6 to 79. It assesses general intelligence through abstract reasoning and problem solving without linguistic, motor or cultural components. It provides a measure of overall intelligence and identifies people with possible intellectual disabilities.
  The test indicates different reference points for the score so that it can be easily interpreted. The reference points are based on the average IQ score (100) and its standard deviation (15). These points are: IQ < 89, indicating that the person is below average; IQ > 111, indicating that the person is above average; 90 > IQ < 110, indicating that the person is average; and finally, IQ >120, indicating that the person is gifted.

CONTACTS AND LOCATIONS:
Overall Officials: Joan Deus-Yela, PhD, Study Director — Universitat Autonoma de Barcelona; Joaquín Ibáñez-Alfonso, PhD, Principal Investigator — Universidad Loyola Andalucia; José Barroso-Tristan, PhD, Principal Investigator — University of Seville
Locations (2):
- Colombia (2):
  - Institución Educativa la Buitrera, Cali, Valle del Cauca Department
  - Colegio Fray Luis Amigo, Cali, Valle del Cauca Department

IPD SHARING:
Plan to Share IPD: No
I do not plan to share the data for ethical, legal, and confidentiality reasons; this clinical data is sensitive, as it pertains to minors.

REFERENCES:
- [Background] Garcia-Navarro C, Company-Cordoba R, Sianes A, Ibanez-Alfonso JA. Cognitive Intervention Programs in Minors Belonging to Disadvantaged Contexts in Spain: A Systematic Review. Children (Basel). 2022 Aug 28;9(9):1306. doi: 10.3390/children9091306. PMID 36138615
- [Background] Ibáñez-Alfonso JA, Company-Córdoba R,, García de la Cadena C. Innovative tools for the assessment of cognitive development in contexts of socioeconomic vulnerability. Practical guide for children and adolescents in Guatemala. 2020
- [Background] Rodriguez-Prieto P, Simpson IC, Gomez-Baya D, Garcia de la Cadena C, Ruiz-Aranda D, Ibanez-Alfonso JA. Neuropsychological Stimulation Program for Children from Low Socioeconomic Backgrounds: Study Protocol for a Randomized Controlled Trial. Healthcare (Basel). 2024 Mar 6;12(5):596. doi: 10.3390/healthcare12050596. PMID 38470707
- [Background] Rodriguez-Prieto P, Giral-Oliveros NA, Simpson IC, Ibanez-Alfonso JA. Cognitive stimulation in socioeconomically disadvantaged children with neurodevelopmental disorders: a case series. Front Psychol. 2024 Jul 9;15:1365697. doi: 10.3389/fpsyg.2024.1365697. eCollection 2024. PMID 39045438
- [Background] Ibanez-Alfonso JA, Company-Cordoba R, Garcia de la Cadena C, Sianes A, Simpson IC. How Living in Vulnerable Conditions Undermines Cognitive Development: Evidence from the Pediatric Population of Guatemala. Children (Basel). 2021 Jan 29;8(2):90. doi: 10.3390/children8020090. PMID 33572817
- [Background] Company-Cordoba R, Gomez-Baya D, Lopez-Gavino F, Ibanez-Alfonso JA. Mental Health, Quality of Life and Violence Exposure in Low-Socioeconomic Status Children and Adolescents of Guatemala. Int J Environ Res Public Health. 2020 Oct 19;17(20):7620. doi: 10.3390/ijerph17207620. PMID 33086701